CLINICAL TRIAL: NCT02498106
Title: Diet and Aggression: Reducing Aggression Among Chronic Psychiatric Inpatients Through Supplementation of Multivitamins, Minerals and n-3 Fatty Acids
Brief Title: Diet and Aggression: Reducing Aggression Among Chronic Psychiatric Inpatients Through Dietary Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Atrium Innovations (Industry)
Responsible Party: Principal Investigator, Erik J. Giltay, MD, PhD, Erik J. Giltay, MD, PhD, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P14.332; 836031016 (Other Grant/Funding Number: ZonMW); NL51850.058.14 (Registry Identifier: Toetsing online); 5176 (Registry Identifier: NTR)
Record Dates: First submitted 2015-07-09; First posted 2015-07-15 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Psychiatric Hospitalization
Keywords: nutrition; aggression; n-3 fatty acids; psychiatry; inpatients admitted >2 years
MeSH Terms: conditions — Aggression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- nutritional supplement (Active Comparator): 2 Orthica Soft Multi Mini capsules and 1 Orthica Fish EPA Mini capsule per day; duration: 6 months
  Interventions: Dietary Supplement: Orthica Soft Multi Mini and Orthica Fish EPA Mini
- placebo (Placebo Comparator): During 6 months one group receives 3 placebo supplements daily with identical look and feel to Orthica Soft Multi Mini and Orthica Fish EPA Mini
  Interventions: Dietary Supplement: Orthica Soft Multi Mini and Orthica Fish EPA Mini

INTERVENTIONS:
Dietary Supplement: Orthica Soft Multi Mini and Orthica Fish EPA Mini — daily intake of 2 Orthica Soft Multi Mini capsules (containing vitamins [B1, B2, B3, B5, B6, B11, B12, C, D, E, Beta Carotene] and minerals [Iodine, Copper, Selenium, Iron, Zinc, Chrome, Manganese]) and 1 Orthica Fish EPA Mini capsule (containing n-3FA: eicosapentaenic acid [EPA] and docosahexaenic acid [DHA])

SUMMARY:
The overall goal of this study is to investigate whether the daily administration of multivitamins, minerals and n-3 fatty acids will reduce aggression in long-term psychiatric inpatients and will thereby reduce costs of care.

DETAILED DESCRIPTION:
Aggressive incidents are highly prevalent among chronic psychiatric inpatients. Previous studies have demonstrated the potential of multivitamin-, mineral-, and n-3 fatty acids (n-3FA) supplementation to reduce aggression in adolescent and forensic populations. To test the hypothesis that multivitamin-, mineral-, and n-3FA supplementation reduces aggression among chronic psychiatric inpatients, we designed a pragmatic, randomised, double-blind, placebo controlled, multicentre intervention study among psychiatric inpatients residing in long-stay psychiatric wards. During 6 months, one group receives 2 supplements daily from Orthica: one containing vitamins and minerals (vitamins [B1, B2, B3, B5, B6, B11, B12, C, D, E, Beta Carotene; Calcium, Iodine, Copper, Magnesium, Selenium, Iron, Zinc, Potassium, Chrome, Manganese]) and one containing fish fatty acids (n-3FA: eicosapentaenic acid [EPA] and docosahexaenic acid [DHA]) and the other group receives 2 placebo capsules.

The main study parameter is the number of aggressive incidents from baseline (t0) to endpoint (six months post baseline, t3). Patients who wish to participate enter a 2-week run-in phase in which they take 2 placebo capsules daily. After positive evaluation of this run-in phase patients are randomized to the active or the control condition. Participants will then start the daily use of 2 supplement capsules or 2 placebo capsules, which will continue for 6 months. At 3 time points (at baseline [t0] and at 2 and 6 months post-baseline [t2 and t3]), three questionnaires measuring feelings of aggression, quality of life, and psychiatric symptoms will be administered. Also, at t0 and t3 (micro)nutrient status will be determined. Finally, at 4 time points (t0, 2 weeks post baseline [t1], t2 and t3), nursing staff will report on observed levels of aggression and social dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* residing at a facility for long-term psychiatric inpatient care
* age 18 or over

Exclusion Criteria:

* pregnancy
* breastfeeding
* known contra-indication for using the supplements used in this study
* expected discharge or transfer within the next 8 weeks
* current use of dietary supplements and refusal to stop using these for the duration of the study
* failure to complete run-in phase
* contra-indication for the use of pork-gelatin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Number of aggressive incidents | daily for the total duration of the (six-month) intervention period
  The main study parameter is the number of aggressive incidents from baseline (t0) to endpoint (six months post baseline, t3), as registered daily on the ward by nurses using the Dutch version of the Staff Observation Aggression Scale- Revised version (SOAS-R)

SECONDARY OUTCOMES:
Patient feelings of aggression | At 3 points (baseline [t0], 2 months post baseline [t2] and six months post baseline[ t3])
  the Aangepaste Versie van de Agressievragenlijst (AVL-AV, 1), a 12 item self-report questionnaire about feelings of aggression.
Patient quality of life | At 3 points (baseline [t0], 2 months post baseline [t2] and six months post baseline[ t3])
  the World Health Organization Quality of Life Questionnaire (WHO-QL-bref 5), a 26-item observer rated quality of life instrument.
Patient psychiatric symptoms | At 3 points (baseline [t0], 2 months post baseline [t2] and six months post baseline[ t3])
  The verkorte Comprehensive Psychopathological Rating Scale (vCPRS), a 25-item observer rated instrument on affective symptoms, which includes the Montgomery-Åsberg Depression Rating Scale (MADRS).
Observed patient social dysfunction | At 4 points (baseline [t0], 2 weeks post baseline [t1], 2 months post baseline[t2] and six months post baseline [t3])
  Nursing staff will fill in the Social Dysfunction Aggression Scale (SDAS), measuring observed levels of aggression and social dysfunction.

OTHER OUTCOMES:
Patient micronutrient status | At 2 points (baseline [t0] and six months post baseline [t3])
  Blood samples (50cc) will be taken to determine micronutrient status, including Vitamins A, E, B1, B6, B12, D, and folate, total iron, magnesium, and the fatty acid spectrum.

CONTACTS AND LOCATIONS:
Overall Officials: Erik J. Giltay, MD PhD, Principal Investigator — Leiden University Medical Center
Locations (6):
- Netherlands (6):
  - GGZ Centraal, Ermelo, Gelderland
  - GGZ Eindhoven, Eindhoven, Noord-Braband
  - GGZ Delfland, Delft, South Holland
  - Fivoor, Den Dolder, Utrecht
  - Rivierduinen, Oegstgeest
  - Parnassia, The Hague

REFERENCES:
- [Background] Hornsveld RH, Muris P, Kraaimaat FW, Meesters C. Psychometric properties of the aggression questionnaire in Dutch violent forensic psychiatric patients and secondary vocational students. Assessment. 2009 Jun;16(2):181-92. doi: 10.1177/1073191108325894. Epub 2008 Oct 13. PMID 18852480
- [Background] Nijman H, Palmstierna T. Measuring aggression with the staff observation aggression scale--revised. Acta Psychiatr Scand Suppl. 2002;(412):101-2. doi: 10.1034/j.1600-0447.106.s412.21.x. PMID 12072137
- [Background] Asberg M, Schalling D. Construction of a new psychiatric rating instrument, the Comprehensive Psychopathological Rating Scale (CPRS). Prog Neuropsychopharmacol. 1979;3(4):405-12. doi: 10.1016/0364-7722(79)90055-9. PMID 400996
- [Background] Skevington SM, Lotfy M, O'Connell KA; WHOQOL Group. The World Health Organization's WHOQOL-BREF quality of life assessment: psychometric properties and results of the international field trial. A report from the WHOQOL group. Qual Life Res. 2004 Mar;13(2):299-310. doi: 10.1023/B:QURE.0000018486.91360.00. PMID 15085902
- [Background] Schoenthaler SJ, Bier ID. The effect of vitamin-mineral supplementation on juvenile delinquency among American schoolchildren: a randomized, double-blind placebo-controlled trial. J Altern Complement Med. 2000 Feb;6(1):7-17. doi: 10.1089/acm.2000.6.7. PMID 10706231
- [Background] Gesch CB, Hammond SM, Hampson SE, Eves A, Crowder MJ. Influence of supplementary vitamins, minerals and essential fatty acids on the antisocial behaviour of young adult prisoners. Randomised, placebo-controlled trial. Br J Psychiatry. 2002 Jul;181:22-8. doi: 10.1192/bjp.181.1.22. PMID 12091259
- [Background] Zaalberg A, Nijman H, Bulten E, Stroosma L, van der Staak C. Effects of nutritional supplements on aggression, rule-breaking, and psychopathology among young adult prisoners. Aggress Behav. 2010 Mar-Apr;36(2):117-26. doi: 10.1002/ab.20335. PMID 20014286
- [Background] Legare N, Brosseau E, Joyal CC. Omega-3 and violence in schizophrenia. Schizophr Res. 2007 Nov;96(1-3):269. doi: 10.1016/j.schres.2007.05.023. Epub 2007 Jul 16. No abstract available. PMID 17629678
- [Background] Benton D. The impact of diet on anti-social, violent and criminal behaviour. Neurosci Biobehav Rev. 2007;31(5):752-74. doi: 10.1016/j.neubiorev.2007.02.002. Epub 2007 Mar 4. PMID 17433442
- [Derived] de Bles NJ, Gast DAA, van der Slot AJC, Didden R, van Hemert AM, Rius-Ottenheim N, Giltay EJ. Lessons learned from two clinical trials on nutritional supplements to reduce aggressive behaviour. J Eval Clin Pract. 2022 Aug;28(4):607-614. doi: 10.1111/jep.13653. Epub 2022 Jan 17. PMID 35040231